CLINICAL TRIAL: NCT00411541
Title: Pulses of Vincristine and Dexamethasone During Maintenance in BFM Protocols for Children With Intermediate-Risk Acute Lymphoblastic Leukemia
Brief Title: Pulses of Vincristine and Dexamethasone in BFM Protocols for Children With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International BFM Study Group (Network)
Collaborators: Associazione Italiana Ematologia Oncologia Pediatrica (Other); BFM-A, Austria (Unknown); BFM-G, Germany and Switzerland (Unknown); CPH, Czech republic (Unknown); European Organisation for Research and Treatment of Cancer - EORTC (Network); Group for Acute Leukemia Treatment (GATLA). (Other); H-POG (Hungary Pediatric Oncology Group) (Other); PINDA, Chile (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-BFM-SG IR ALL
Record Dates: First submitted 2006-12-13; First posted 2006-12-14 (Estimated); Last update posted 2006-12-14 (Estimated); Status verified 2006-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: acute lymphoblastic leukemia, maintenance, BFM protocol; intermediate risk childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine; Dexamethasone

INTERVENTIONS:
Drug: vincristine
Drug: dexamethasone

SUMMARY:
Studies in the 1970s and 1980s suggested that the outcome of childhood acute lymphoblastic leukemia could be improved by intensification of conventional continuation chemotherapy with pulses of vincristine sulfate and steroids. We aimed to investigate the efficacy and toxic effects of vincristine-dexamethasone pulses as an addition to the continuation-therapy phase in a large cohort of children with intermediate-risk disease who were treated with the BFM treatment strategy

DETAILED DESCRIPTION:
The study enrols children from 8 participating organizations. All children are treated with similar protocols based on the BFM treatment strategy, which include induction, consolidation, reinduction and continuation-therapy phases. At the beginning of the continuation-therapy phase, those patients in complete remission are randomly assigned to either a treatment or a control group. Control patients are given conventional mercaptopurine and methotrexate chemotherapy only. Patients in the treatment arm are also given pulses of vincristine (1.5 mg/sqm weekly for 2 weeks) and dexamethasone (6 mg/sqm daily for 7 days) every 10 weeks for six cycles.

ELIGIBILITY:
Inclusion Criteria:

* age <1 or >5 years or
* white blood cell count at diagnosis >=20000

Exclusion Criteria:

* prednisone poor response
* no complete remission at the end of induction (IA)
* t(9,22) clonal translocation
* t(4,11) clonal translocation

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2600
Dates: Start 1995-04; Study Completion 2004-01

PRIMARY OUTCOMES:
disease free survival

SECONDARY OUTCOMES:
survival

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schrappe, MD, Principal Investigator — BFM-G, Germany and Switzerland; Helmut Gadner, MD, Principal Investigator — BFM-A, Austria; Giuseppe Masera, MD, Principal Investigator — AIEOP, Itlay; Jan Stary, MD, Principal Investigator — CPH, Czech republic; Ives Benoit, MD, Principal Investigator — EORTC-CLG, France, Belgium, Portugal; Edina Magyarosy, MD, Principal Investigator — H-POG (Hungary Pediatric Oncology Group); Myriam Campbell, MD, Principal Investigator — PINDA, Chile; Eduardo Dibar, MD, Principal Investigator — Group for Acute Leukemia Treatment (GATLA).
Locations (8):
- Department of Pediatric Hematology-Oncology, Italian Hospital, Buenos Aires, Argentina
- Children's Cancer Research Institute, St Anna Kinderspital, Vienna, Austria
- Department of Pediatric Hemato-Oncology, Gent University Hospital, Ghent, Belgium
- Department of Pediatrics Hematology and Oncology, Hospital Roberto del Rio, Santiago, Chile
- Department of Pediatric Hematology and Oncology, University Hospital Motol, Prague, Czechia
- Medizinische Hochschule Hannover, Hanover, Germany
- Department of Pediatrics, Semmelweis University, Budapest, Hungary
- Pediatric Clinic - University of Milano-Bicocca, Monza, Italy

REFERENCES:
- [Derived] Conter V, Valsecchi MG, Silvestri D, Campbell M, Dibar E, Magyarosy E, Gadner H, Stary J, Benoit Y, Zimmermann M, Reiter A, Riehm H, Masera G, Schrappe M. Pulses of vincristine and dexamethasone in addition to intensive chemotherapy for children with intermediate-risk acute lymphoblastic leukaemia: a multicentre randomised trial. Lancet. 2007 Jan 13;369(9556):123-31. doi: 10.1016/S0140-6736(07)60073-7. PMID 17223475